CLINICAL TRIAL: NCT02972294
Title: HiFIT Study: Interest of Intravenous Iron and Tranexamic Acid to Reduce Transfusion in Hip Fracture Patients
Brief Title: HiFIT Study : Hip Fracture: Iron and Tranexamic Acid
Acronym: HiFIT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 1year inclusion hold due to PV new fact (Monofer hold for risk revaluation) DSMB Interim analysis : 1treatment with important transfusion risk reduction/inclusions issues (COVID)/sites change of practice if study continue=>stop inclusions
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 49RC16_0014
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Hip Fractures Pathologic; Anemia
Keywords: iron isomaltoside; tranexamic acid
MeSH Terms: conditions — Anemia | interventions — iron isomaltoside 1000; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TXA + IIM (Experimental): The patients randomized to this arm will have iron isomaltoside 1000 and tranexamic acid
  Interventions: Drug: Iron Isomaltoside 1000; Drug: Tranexamic Acid
- Placebo TXA + IIM (Experimental): The patients randomized to this arm will have iron isomaltoside 1000 and Placebos tranexamic acid
  Interventions: Drug: Iron Isomaltoside 1000; Drug: Placebos tranexamic acid
- TXA + Placebo IIM (Experimental): The patients randomized to this arm will have Placebos iron isomaltoside 1000 and tranexamic acid
  Interventions: Drug: Tranexamic Acid; Drug: Placebos iron isomaltoside 1000
- Placebo TXA + Placebo IIM (Experimental): The patients randomized to this arm will have Placebos iron isomaltoside 1000 and Placebos tranexamic acid
  Interventions: Drug: Placebos iron isomaltoside 1000; Drug: Placebos tranexamic acid

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — Iron Isomaltoside 1000 will be use. Blinding procedure will be put in place for the administration of the treatment
  Other Names: monofer
  Arms: Placebo TXA + IIM; TXA + IIM
Drug: Tranexamic Acid — Tranexamic acid will be use.
  Other Names: exacyl
  Arms: TXA + IIM; TXA + Placebo IIM
Drug: Placebos iron isomaltoside 1000 — placebo of Iron Isomaltoside 1000 correspond to a saline solution. Blinding procedure will be put in place for the administration of this treatment
  Other Names: saline serum
  Arms: Placebo TXA + Placebo IIM; TXA + Placebo IIM
Drug: Placebos tranexamic acid — placebo of tranexamic acid correspond to a saline solution.
  Other Names: saline serum
  Arms: Placebo TXA + IIM; Placebo TXA + Placebo IIM

SUMMARY:
Fractures of the upper end of the femur, called commonly "Hip fractures" are very common, with an incidence of approximately 1.6 million cases per year worldwide. This high incidence is anticipated to grow rapidly in the next decades, driven by population aging. Anemia is very frequent on admission for hip fracture, concerning up to 45% of the patients, with a mean hemoglobin level of 12.5±0.2 g/dl. This high prevalence of anemia together with blood losses, secondary to the fracture itself and surgery are responsible for a high rate of blood transfusion (approximately 40-50% of the patients). However, both anemia and blood transfusion are associated with poor outcome, including increased mortality, length of stay, infection rate etc. In addition, blood is a scarce and expensive resource and its use should be limited as much as possible. There is therefore a need to treat this anemia and/or to prevent the decrease in hemoglobin. For this purpose, intravenous iron has been proposed. Some non-randomized, mainly retrospective, studies have shown that perioperative intravenous iron was able to reduce blood transfusion (i.e. the number of patients transfused and the number of units per patient). Another way to reduce blood transfusion would be to reduce perioperative bleeding. Tranexamic acid has proven to be efficient for this purpose both in trauma patients and in elective surgery patients.The interest for perioperative blood management has recently increased thanks to better recognition of the adverse effects of blood transfusion, better understanding of iron metabolism, new intravenous iron drugs and a renewed interest in former medications (i.e. tranexamic acid). HiFIT study therefore propose a 2X2 factorial design for this study in order to answer questions vis-à-vis the interest of iron and tranexamic acid to reduce blood transfusion in hip fracture patients.

DETAILED DESCRIPTION:
Fractures of the upper end of the femur, called commonly "Hip fractures"are very common, with an incidence of approximately 1.6 million cases per year worldwide. This high incidence is anticipated to grow rapidly in the next decades, driven by population aging. Anemia is very frequent on admission for hip fracture, concerning up to 45% of the patients, with a mean hemoglobin level of 12.5±0.2 g/dl. This high prevalence of anemia together with blood losses, secondary to the fracture itself and surgery are responsible for a high rate of blood transfusion (approximately 40-50% of the patients). However, both anemia and blood transfusion are associated with poor outcome, including increased mortality, length of stay, infection rate etc. In addition, blood is a scarce and expensive resource and its use should be limited as much as possible. There is therefore a need to treat this anemia and/or to prevent the decrease in hemoglobin. For this purpose, intravenous iron has been proposed. Some non-randomized, mainly retrospective, studies have shown that perioperative intravenous iron was able to reduce blood transfusion (i.e. the number of patients transfused and the number of units per patient). Indeed, a pooled analysis of 5 studies including 1,361 patients suggests that intravenous iron could reduce perioperative transfusion in hip fracture patients. However, there is no definitive data. Another way to reduce blood transfusion would be to reduce perioperative bleeding. Tranexamic acid has proven to be efficient for this purpose both in trauma patients and in elective surgery patients. However, there are only two randomized studies investigating the interest of tranexamic acid in hip fractures, and they are not conclusive probably owing to a lack of power. In addition, use of intravenous tranexamic acid could be limited in this population of frail patients and topical use of tranexamic acid, notably to prevent the intraoperative bleeding, appear to be an accurate and sure alternative.

Although hip fracture is a very frequent pathology, with a high burden of care, few data are available that focus on the management of perioperative anemia in this context. The interest for perioperative blood management has recently increased thanks to better recognition of the adverse effects of blood transfusion, better understanding of iron metabolism, new intravenous iron drugs and a renewed interest in former medications (i.e. tranexamic acid). hiFIT study therefore propose a 2X2 factorial design for this study in order to answer questions vis-à-vis the interest of iron and tranexamic acid to reduce blood transfusion in hip fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Osteoporotic Fractures of the upper end of the femur requiring surgical repair.
* Preoperative hemoglobin between 9.5 and 13 g/dl.
* Patient or relative signed informed consent or inclusion thanks to urgent inclusion procedure

Exclusion Criteria:

* Bone marrow disease or ongoing treatment (such as chemotherapy), which could interfere with bone marrow erythropoiesis,
* Known allergy or counter-indication to iron and/or to tranexamic acid,
* Uncontrolled arterial hypertension,
* Recent iron infusion (within one week),
* Blood transfusion within one week before inclusion or preoperative blood transfusion already scheduled,
* Any patient who cannot be transfused or has refused consent for a blood transfusion,
* Bedridden or very dependent patient (equivalent to GIR 1 or 2 class).
* Non-affiliation to French health care coverage,
* Adult patient protected under the law (guardianship),
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who received a blood transfusion during their hospital stay following surgery | From the day of surgery until hospital discharge (or until day 30 if patient is still hospitalized).
  Proportion of patients who received a blood transfusion during their hospital stay following surgery

SECONDARY OUTCOMES:
Proportion of patients who received a blood transfusion after surgery | From the day of surgery until Day 3, Day 7 and Day 30 post surgery.
  Proportion of patients who received a blood transfusion during the month following surgery (including fresh frozen plasma and platelets)
Number of packed red blood cell units transfused per patient, as well as number of fresh frozen plasma and platelets units | Till postoperative Day3, first week posteratively,and till hospital discharge (or one month if patients still hospitalised)
  Number of packed red blood cell units transfused per patient, as well as number of fresh frozen plasma and platelets units
Hemoglobin concentration | At inclusion and on days 3, 7 (or hospital discharge if it happens first) and 30.
  Hemoglobin concentration
Proportion of patients with anemia (hemoglobin <12 g/dL in women and <13 g/dL in men) | At inclusion and on days 3, 7, hospital discharge (if it happens before Day 30) and 30.
  Proportion of patients with anemia (hemoglobin <12 g/dL in women and <13 g/dL in men)
Reticulocytes count | On days 3, 7 (or hospital discharge if it happens first) and 30 post surgery
  Reticulocytes count
Perioperative blood loss (estimated according to a formula based on hematocrit variation). | During surgery
  Perioperative blood loss (estimated according to a formula based on hematocrit variation): (HtD0 - HtD3)*TBV + number of RPBC transfused unit x 200 ml. Ht = Haematocrit, TBV = total blood volume (70 mL/kg in men and 65 mL/kg in women)
Post operative Iron deficiency rate | On Day 7 (or hospital discharge if it happens first) and Day 30.
  Proportion of patients with Iron deficiency (defined as a ferritin < 100 ng/ml or < 300 ng/ml together with transferrin saturation <20%), measurement of ferritin and transferrin saturation
Number of hospitalization days | On Day 30 and Day 90 following surgery.
  Number of hospitalization days
Proportion of patients at home | On Day 30 and Day 90.
  Proportion of patients returned at home (or at their previous place of living)
Proportion of patients able to walk a distance of ten feet without assistance | On Day 30 and Day 90
  Proportion of patients able to walk a distance of ten feet without assistance
Variation of quality of life | From inclusion to Day 30 and Day 90
  Variation of EQ-5D score
Variation of perceived quality of life | From inclusion to Day 7 (or hospital discharge if it happens first) and Day 90.
  Variation of perceived quality of life with a single overall item from PQOL scale
Variation of IADL test | From inclusion to Day 90.
  Variation of IADL test
Death rate from all causes | From inclusion to Day 90
  Death rate from all causes
Rate of adverse events including the following clinical complications: Vascular events, Heart failure; Renal failure; Infectious complications; Anaphylactic reaction; Transfusion-related complications | From inclusion to Day 90
  Rate of adverse events including the following clinical complications: Vascular events, Heart failure; Renal failure; Infectious complications; Anaphylactic reaction; Transfusion-related complications

OTHER OUTCOMES:
Strength assessed by the Hand Grip Strength test | On day 7 (or hospital discharge if it happens first)
  Maximum strength of the hand and forearm muscles assessed by the Hand Grip Strength test
Muscular fatigability assessed by the Hand Grip Strength test | On day 7 (or hospital discharge if it happens first)
  Muscular fatigability between the first attempt and the third attempt of the Hand Grip Strength test (variation of the maximum strength measured at the first and the third atempt)
Level of locomotion and balance assessed by the Timed " Up and Go " test. | On day 7 (or hospital discharge if it happens first)
  Level of locomotion and balance assessed by the Timed " Up and Go " test,

CONTACTS AND LOCATIONS:
Overall Officials: Sigismond SL Lasocki, PU-PH, Study Director — UNIVERSITE HOSPITAL, ANGERS
Locations (13):
- France (13):
  - CHU Angers - DEPARTEMENT D'ANESTHESIE REANIMATION, Angers
  - Clinique de L'Anjou- Anesthesie Reanimation, Angers
  - HIA Clermont-Tonnerre, Brest
  - Chu Grenoble - Departement D'Anesthesie Reanimation, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHU Lille, Lille
  - Hospices Civils Lyon, Lyon
  - Ramsay Santé, Clinique de la Sauvegarde, Lyon
  - Chu Montpellier - Departement D'Anesthesie Reanimation, Montpellier
  - Chu Nantes- Service de Reanimation Chirurgicale, Nantes
  - Chu Poitiers - Service D'Anesthesie Reanimation, Poitiers
  - Chu Rennes - Service D'Anesthesie Reanimation, Rennes
  - Medipôle, Villeurbanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lasocki S, Capdevila X, Bijok B, Lahlou-Casulli M, Collange V, Grillot N, Loupec T, Rineau E, Leger M; HiFIT Investigators. Quality of life of patients with hip fracture was better during the COVID-19 period than before, an ancillary study from the HiFIT multicenter study. Front Public Health. 2024 Apr 16;12:1362240. doi: 10.3389/fpubh.2024.1362240. eCollection 2024. PMID 38689774
- [Derived] Lasocki S, Capdevila X, Vielle B, Bijok B, Lahlou-Casulli M, Collange V, Grillot N, Danguy des Deserts M, Duchalais A, Delannoy B, Drugeon B, Bouzat P, David JS, Rony L, Loupec T, Leger M, Rineau E; HiFIT Investigators; SFAR research network. Ferric derisomaltose and tranexamic acid, combined or alone, for reducing blood transfusion in patients with hip fracture (the HiFIT trial): a multicentre, 2 x 2 factorial, randomised, double-blind, controlled trial. Lancet Haematol. 2023 Sep;10(9):e747-e755. doi: 10.1016/S2352-3026(23)00163-1. Epub 2023 Jul 28. PMID 37524101
- [Derived] Lasocki S, Bruckert V, Campfort M, Leger M, Rineau E. Restrictive transfusion targets the heart now! Insight from the REALITY study. Anaesth Crit Care Pain Med. 2021 Apr;40(2):100854. doi: 10.1016/j.accpm.2021.100854. Epub 2021 Mar 27. No abstract available. PMID 33781988
- [Derived] Lasocki S, Loupec T, Parot-Schinkel E, Vielle B, Danguy des Deserts M, Roquilly A, Lahlou-Casulli M, Collange V, Desebbe O, Duchalais A, Drugeon B, Bouzat P, Garrigue D, Mounet B, Hamard F, David JS, Leger M, Rineau E; HiFIT Study Group. Study protocol for a multicentre, 2x2 factorial, randomised, controlled trial evaluating the interest of intravenous iron and tranexamic acid to reduce blood transfusion in hip fracture patients (the HiFIT study). BMJ Open. 2021 Jan 17;11(1):e040273. doi: 10.1136/bmjopen-2020-040273. PMID 33455926